CLINICAL TRIAL: NCT03852901
Title: Sodium-Glucose CoTransporter 2 (sGLT2) Inhibitor and Endogenous Ketone Production
Brief Title: Sodium-glucose Co Transporter 2 (sGLT2) Inhibitor and Endogenous Ketone Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190060; 19-AG-0060
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-12-13

CONDITIONS: Empaglifozin; Physiological Effects of Drugs; Hypoglycemic Agents; Sodium-Glucose Transporter 2 Inhibitors
Keywords: Ketones; Metabolism; Hormones; Alzheimer's Disease
MeSH Terms: conditions — Ketosis; Alzheimer Disease | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single group
  Interventions: Drug: empagliflozin (Jardiance) 25 mg

INTERVENTIONS:
Drug: empagliflozin (Jardiance) 25 mg — Oral empagliflozin 25 mg/day x 14 days

SUMMARY:
Background:

The drug empagliflozin treats diabetes. It lowers blood sugar by increasing glucose the kidneys excrete. This increases levels of ketones formed in the blood. The body makes ketones when it does not have enough glucose for fuel. The brains of many people with age-related diseases like Alzheimer's do not use glucose well. Brain use of ketones might improve mental ability. We investigated how empagliflozin affects ketone levels, which could lead to ways to improve brain health as people age.

Objectives:

To study how taking empagliflozin affects systemic and brain metabolism including ketone levels in people without diabetes.

Eligibility:

Adults at least 55 years old without diabetes

Design:

After a screening Visit, eligible participants were admitted to the NIA Clinical Unit during Visits 1 (baseline), 2 (first dose) and 3 (last/14th dose). On each Visit, blood draws were performed and circulating metabolites and hormones were repeatedly measured over 34-hour periods. Using plasma from fasting state only, we isolated total and neuronal-origin extracellular vesicles to measure proteins of the IGF-1 and insulin signaling cascades. Furthermore, on each Visit, we performed magnetic resonance spectroscopy (MRS) to measure concentrations of a plethora of metabolites in the brain. Between Visits 2 and 3, participants were taking the drug at home. A continuous glucose monitoring device was placed to detect potential glucose fluctuations while at home. The study was concluded for participants after the end of Visit 3.

DETAILED DESCRIPTION:
Objective and Specific Aims: The objective of this proof-of-concept study was to demonstrate in non-diabetic men and women age > 55 years that a sGLT2 inhibitor (empagliflozin) can increase ketone bodies and metabolites used for gluconeogenesis. We also hypothesized that empagliflozin would increase circulating glucagon and fatty acids, decrease circulating amino acids, upregulate IGF-1 and insulin cascades in plasma extracellular vesicles, and change MRS brain metabolism measures.

Experimental Design and Methods: men and women (total n=21) were recruited for this pilot study. Each eligible participant had a screen visit (Visit 0) and three additional 2-day study visits (Visit 1-3). On Visits 1, 2 and 3, frequent blood sampling for beta-hydroxybutyrate butyrate (BHB), acetoacetate (AcAc), fatty and amino acids, glucagon, insulin and glucose levels will be carried out; these visits also included blood work for extracellular vesicle biomarkers and brain MRS. In addition, placement of a continuous glucose monitor (CGM) along with a 34-hour urine collection was carried out. On Visit 2 the participants wore the CGM until they returned for their next Visit. On Visit 3 the CGM was removed at the end of the study Visit. On Visit 1, no empagliflozin was administered. Participants returned in 13 +/- 2 days for Visit 2. Visit 2 was the same as Visit 1 except empagliflozin 25 mg was administered both mornings, at least 30 minutes before eating breakfast and participants continueed empagliflozin 25 mg once every morning, at least 30 minutes before eating breakfast, at home until they returned in 13 +/- 2 days for Visit 3. At the end of Visit 3, empagliflozin was stopped.

Medical Relevance and Expected Outcome: Elevating ketone bodies may bolster neuronal health and delay onset and progression of cognitive impairment. The expected outcome of this study was an increase in circulating levels of ketones, glucagon and fatty acids, an increased expression of receptors and mediators of ketone metabolism in plasma exosomes, an upregulation of IGF-1/insulin cascades in exosomes, and a change in Magnetic Resonance Spectroscopy (MRS) brain metabolism measures, in subjects taking a sGLT2 inhibitor. We expected circulating amino acid levels to decrease, especially during the overnight hours. This study will aid in deciding whether this class of compound may be used in a larger study to improve cognitive function in patients with diagnosis consistent with declining cognitive function. We required that empagliflozin was taken for up to 2 weeks before returning for Visit 3, because we needed to fully understand the homeostatic adaptations that may occur in the metabolite response to empagliflozin due to prolonged (up to 2 weeks) sGLT2 inhibition. It is our goal in the future to use the information gathered in this pilot study to design a long-term study in people who actually suffer from mild cognitive impairment/Alzheimer's disease and therefore a Visit 2 (34-hour acute study) only, as outlined above, would not give us the full picture of the metabolic changes that might occur with prolonged use, especially in a non-diabetic population.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 55 years and older.
* Healthy (see exclusion criteria below).
* Able to understand the study risks and procedures, and consent to participate in the study.
* Able to read and speak English.

EXCLUSION CRITERIA:

* History of diabetes (requiring any medical treatment other than diet and exercise) or fasting plasma glucose > 126 mg/dl or HbA1c> 6.5 %.
* History of hypoglycemia.
* BMI > 35 kg/m(2).
* Creatinine clearance less than 60 ml/min as measured by GFR.
* Glucosuria
* History of anemia within the past 6 months or Hgb <11.0 mg/dL for women and Hgb <12.5 mg/dL for men.
* Current steroid use or steroid use within 90 days of screening, excluding eye drops.
* Currently taking loop diuretics (Lasix, for example).
* Participant presently following a calorie restriction diet, low carb/high fat diet.
* HIV virus infection
* Hepatitis B infection, as evidenced by a positive HBsAG at screen visit.
* Hepatitis C infection that has not been treated. (The screen blood work must show HCV RNA quantitative is not detectable).
* Active infection/fever that may cause changes in glucose metabolism.
* Known allergy to sGLT2 inhibitors in the past.
* Thyroid dysfunction that is not controlled or treated. This will be determined by Free T3, T4, Free T4 or TSH not within MedStar Harbor Hospital laboratory normal ranges for this pilot study.
* Adrenal dysfunction as determined by a cortisol level not within the normal range for MedStar Harbor Hospital Laboratory for this pilot study.
* Kidney or liver disease, (GFR < 60 mL/min/1.73 m(2) and/or liver enzymes not within normal ranges for MedStar Harbor Hospital Laboratory for this pilot study.
* Severe gastrointestinal diseases such as Crohn s disease or ulcerative colitis requiring continuous treatment.
* History of severe pulmonary disease such as chronic obstructive pulmonary disease (COPD) or asthma requiring continuous medication use.
* Patients with known, or evidence of, peripheral vascular disease.
* History of chronic urinary tract infections.
* History of recurrent or recent dehydration in the past year.
* History of recurrent or recent vaginal yeast infection.
* Alcohol intake greater than 30 grams (drink more than 2 beers OR equivalent per day).
* History of severe psychiatric conditions associated with behavioral problems or requiring chronic medical treatment.
* Poor venous access.
* Inability to walk 2,000 steps
* Donation or loss of 400 mL or more of blood within 56 days prior to and subsequent to screening.
* Participation in another study in the past 30 days, in which a study drug was administered.
* Currently participating in another study unless the investigator feels it would not interfere with the study.
* History of a medical condition or any other reason that, in the opinion of the investigator, will make participation in this study unsafe.
* Blood work or urine tests that are not considered by the study physician to be in an acceptable range for the study.
* Metal implants and devices incompatible with 3T Magnetic Resonance Imaging (MRI), or another contraindication to MRI.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-AG-0060.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: The single group of the study (empagliflozin group) took empagliflozin 25mg/day for 14 days.
Period: Overall Study
Arm/Group | Single Arm
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: The single group underwent baseline assessment (visit 1). Fourteen days later (visit 2), participants took the first empagliflozin dose and acute effects were assessed. Participants continued taking empagliflozin once per day at home for 13 additional days, and returned for the final visit (visit 3) in which chronic effects were assessed.
Arm/Group | Single Arm
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.14 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum β-hydroxybutyrate (BHB)
Description: Change in serum β-hydroxybutyrate (BHB) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: µM
Arm/Group | Single Arm
Number analyzed (Participants) | 21
µM | 40.717 (4.866)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p < 0.001, Mixed Models Analysis — Type III of fixed effects. Num df = 1; Den df = 902.758; F = 70.003; Sig. < 0.001 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit & Timepoint; Fixed effects: Visit, Timepoint, Sex, Visit*Sex; Mean Difference (Final Values) = 40.717, 95% CI 2-sided [31.166 to 50.268], Standard Error of Mean 4.866

2. Secondary Outcome: Change in Plasma Glucose
Description: Change in plasma glucose after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Single Arm
Number analyzed (Participants) | 21
mg/dl | -.637 (1.051)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.545, Mixed Models Analysis — Type III of fixed effects. Num df = 1; Den df = 884.229; F = .367; Sig = .545 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit & Timepoint; Fixed effects: Visit, Timepoint, Sex, Visit*Sex; Mean Difference (Final Values) = -0.637, 95% CI 2-sided [-2.699 to 1.426], Standard Error of Mean 1.051

3. Secondary Outcome: Change in Serum Non-esterified Fatty Acids (NEFAs)
Description: Change in serum non-esterified fatty acids (NEFAs) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | Single Arm
Number analyzed (Participants) | 21
mEq/L | .027 (.009)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.003, Mixed Models Analysis — Type III of fixed effects. Num df = 1; Den df = 880.629; F = 8.782; Sig. = 0.003 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit & Timepoint; Fixed effects: Visit, Timepoint, Sex, Visit*Sex; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [.009 to .044], Standard Error of Mean .009

4. Secondary Outcome: Change in Plasma Insulin
Description: Change in plasma insulin after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mIU/L
Arm/Group | Single Arm
Number analyzed (Participants) | 21
mIU/L | -2.647 (1.329)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.047, Mixed Models Analysis — Type III of fixed effects. Num df = 1; Den df = 880.870; F = 3.970; Sig. = 0.047 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit & Timepoint; Fixed effects: Visit, Timepoint, Sex, Visit*Sex; Mean Difference (Final Values) = -2.647, 95% CI 2-sided [-5.255 to -0.040], Standard Error of Mean 1.329

5. Secondary Outcome: Change in Serum Acetoacetate (AcAc)
Description: Change in serum Acetoacetate (AcAc) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: µM
Arm/Group | Single Arm
Number analyzed (Participants) | 21
µM | -5.573 (1.853)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.003, Mixed Models Analysis — Type III of fixed effects. Num df = 1; Den df = 902.181; F = 9.049; Sig. = 0.003 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit & Timepoint; Fixed effects: repeated-measures. Visit, Timepoint, Sex, Visit*Sex; Mean Difference (Final Values) = -5.573, 95% CI 2-sided [-9.210 to -1.937], Standard Error of Mean 1.853

6. Secondary Outcome: Change in 1H MRS BHB
Description: Change in 1H MRS β-hydroxybutyrate (BHB) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Single Arm
Number analyzed (Participants) | 20
mmol/L | 0.04 (0.03)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.5849, Mixed Models Analysis — Type III of fixed effects. Num df: 2; Den df = 33; F = 0.5451; Sig. = 0.5849 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit; Fixed effects: Visit, Sex, Age, fCSF

7. Secondary Outcome: Change in 1H MRS Glutamate (Glu)
Description: Change in 1H MRS glutamate (Glu) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Single Arm
Number analyzed (Participants) | 20
mmol/L | -0.23 (0.11)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.0142, Mixed Models Analysis — Type III of fixed effects. Num df = 2; Den df = 35; F = 4.8191; Sig. = 0.0142 (threshold for statistical significance p < 0.05); Random effect: ID; Repeated measures: Visit; Fixed effects: Visit, Sex, Age, fCSF

8. Secondary Outcome: Change in 1H MRS Glutamine (Gln)
Description: Change in 1H MRS glutamine (Gln) after 14 days on empagliflozin, compared with baseline.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Single Arm
Number analyzed (Participants) | 20
mmol/L | -0.27 (0.12)
Statistical Analysis 1: Comparison: Single Arm; No a-priori power calculation was performed due to the exploratory nature of the study; Test type: Other; p = 0.024, Mixed Models Analysis — Type III of fixed effects. Num df: 2; Den df = 34; F = 4.1501; Sig. = 0.0244 (threshold for statistical significance p < 0.05); Random effects: ID; Repeated measures: Visit; Fixed effects: Visit, Sex, Age and fCSF

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=21)
Mild creatinine elevation (Renal and urinary disorders) | 1 (1) — Mild creatinine elevation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT03852901/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03852901/ICF_001.pdf